CLINICAL TRIAL: NCT04209907
Title: the Effect of Retrolaminar Block on Post Operative Analgesia After Lumbar Vertebra Surgery
Brief Title: the Effect of Retrolaminar Block on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kevser Peker, assitant professor, Kırıkkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: retolaminar block
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group which retrolaminar block will be approved (Active Comparator): the retrolaminar block will be made for postoperative analgesia
  Interventions: Other: retrolaminar block tecnique
- the group which retrolaminar block will not be approved (No Intervention): the retrolaminar block will not be made for postoperative analgesia

INTERVENTIONS:
Other: retrolaminar block tecnique — By using ultrasound probe, the needle with in-plane , after seeing vertebral lamina, the local anesthetic will injectate
  Arms: the group which retrolaminar block will be approved

SUMMARY:
In recent years, as a part of multimodal analgesia, paravertebral blocks are replacing epidural analgesia due to the less side effects. Although the risk of pneumothorax is the most feared complication in paravertebral blocks, retrolaminar block (RLB) -which is a paravertebral block- significantly reduces this risk due to the anatomical technique of procedure. The investigators aim to investigate the effect of retrolaminar block with ultrasound- guided on perioperative analgesia for patients undergoing lumbar vertebra surgery.

DETAILED DESCRIPTION:
Retrolaminar block will applie before general anesthesia induction when patients will be awake and under midazolam (0.03 mg/kg) sedation and standardized monitoring at the preoperative block area in sitting position using in-plane approach. After sterilising the skin, the investigators will perform block by using 7-18 MHz convex ultrasound probe ( Esaote My Lab 6 US Machine, Florance, Italy) and a 22-gauge, 100-mm Stimuplex needle (B. Braun, Germany). The investigators will pass in a sagittal plane from medial to lateral at the mid-lomber level, and identified the hyperechoic laminae, transverse processes, ribs and pleura.

The L3 laminae will be identified approximately lateral of the spinous process. The needle will insert in-plane, cephalad to caudad. After lamina contact and negative aspiration, 20 ml bupivacaine 0.25% will be injected at low pressure with intermittent negative aspiration on each side and spread of local anesthetic between laminae and paraspinous muscles will be seen without pain or paresthesia. Then 30 minutes later, the patient will be taken to the operating room.

After general anesthesia prosedure, the patients will evaluate whether they have pain throughout 24 hours after the operation. The pain scores will be evaluated with visuel analogue scale.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old
2. ASA 1, 2, 3 patients
3. undergoing lumvar vertyebra surgery

Exclusion Criteria:

1. pregnant woman
2. child
3. patint wiht cognitive disfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
change of pain throughout postoperative 24 hours | change in postoperative 24 hours
  visuel analogue scale is used for post operative pain evaluation. it is range from 0 to 10. 0 is used for no pain, 10 is used severe pain. the investigors will evaluate the postoperative pain with visuel analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Peker, Principal Investigator — Kırıkkale University Faculty of Medicine
Locations (1):
- Kırıkkale Univercity Faculty of Medicine Hospital, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peker K, Aydin G, Gencay I, Saracoglu AG, Sahin AT, Ogden M, Peker SA. The effect of preemptive retrolaminar block on lumbar spinal decompression surgery. Eur Spine J. 2024 Nov;33(11):4253-4261. doi: 10.1007/s00586-024-08219-4. Epub 2024 Jun 17. PMID 38886235